CLINICAL TRIAL: NCT03278366
Title: The Effects of Dance Practice on Assessment Score Performance, Behavior and Attendance in a Public School District With High Rates of Economically Disadvantaged Elementary Students.
Brief Title: Effects of Dance Practice in Elementary Students
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Suspended secondary to COVID-19 and decreased access to school setting
Sponsor: Skidmore College (Other)
Responsible Party: Principal Investigator, Sarah DiPasquale, Assistant Professor, Skidmore College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1704-605
Record Dates: First submitted 2017-08-29; First posted 2017-09-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Educational Activities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dancing students (Experimental): Students will participate in dance activities from a video with their teacher in class.
  Interventions: Behavioral: Dancing
- Non-Dancing Students (No Intervention): Students will continue with typical classroom activities in class and will not participate in dancing activities

INTERVENTIONS:
Behavioral: Dancing — Participants in the intervention group will participate in daily dance activities with their teacher by following along with a video created by the dance researchers at Skidmore College. Teachers will be specifically asked to utilize the movement phrases just prior to administering any formal assessment activity within their classroom (tempo may be chosen at teacher's discretion). Furthermore, teachers may choose to utilize the dance phrases as 'brain breaks' at any point throughout their school day.
  Arms: Dancing students

SUMMARY:
The purpose of this study is to assess changes in benchmark and state assessment scores in a public elementary school following an intervention of dance integration into the daily routine of the classroom. Furthermore, this study aims to assess if dance may improve student behavior, teacher perception of student behavior, reading level and attendance.

DETAILED DESCRIPTION:
The use of movement in primary school classrooms is a longstanding practice drawn upon by teachers in various ways. Dance movement in particular is popular among teachers for several reasons: it is enjoyable for students, it can be imaginative, it engages the body as well as the brain, and it can be made accessible to students of varying abilities.

In the field of education, the use of brief bouts of physical activity (PA) or 'brain breaks' have been gaining attention. Teachers have reported perceived improved student concentration during the academic school day by utilizing PA in both elementary and middle school populations. Carlson et al. suggest that PA breaks can indeed improve overall student behavior in the classroom while Donnelly and Lambourne report a 6% improvement on standardized tests in classrooms incorporating PA into academic lessons. Erwin et al. describe improvements in math and reading fluency standardized test scores following an intervention of PA incorporated into an elementary classroom. More conclusive research is indeed needed, yet incorporating PA into the culture of an academic environment appears to hold some merit.

The US Department of Education alongside the National Dance Education Organization published a paper outlining the research priorities for dance education in 2004.

"Of 20 Issues researched in the Research Dance Education project, 15 Issues were identified as gaps, and are therefore identified as Issues in need of future research…The 15 severely under-researched issues over decades impact policy and pedagogy at state and national levels, specifically: Multicultural Education, Integrated Arts, Policy, Affective Domain, Interdisciplinary Education, Student Achievement, Equity, National Content Standards, Funding, Student Performance, Children at Risk, Certification, Teacher Standards, Uncertified Teachers, and Brain Research."

Despite this call to action over a decade ago, to the investigators knowledge, a study assessing change in academic performance following an intervention of dance in a public school serving students with high rates of economic disadvantage has not been published.

The purpose of this study is to assess changes in benchmark and state assessment scores in a public elementary school following an intervention of dance integration into the daily routine of the classroom. Furthermore, this study aims to assess if dance may improve student behavior, teacher perception of student behavior, reading level and attendance. The investigators hypothesize that positive improvements may be observed in all variables by integrating dance into the academic classroom.

ELIGIBILITY:
Inclusion criteria:

Inclusion criteria:

* Registration in an elementary classroom at Boulevard Elementary school, Gloversville Enlarged School District; Gloversville, New York
* Registration in an elementary classroom Park Terrace Elementary school, Gloversville Enlarged School District; Gloversville, New York
* Participating in a classroom where teacher is utilizing dance integration into their curriculum.

Exclusion Criteria:

• None

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 349 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Benchmark/Summative assessments | Baseline, 8 weeks, 16 weeks, 24 weeks.
  Unit/chapter assessments in Math and English Language Arts
Change in State Assessment scores | Baseline and 9 months.
Attendance/tardiness | 10 months.
  Student attendance
Change in Reading Level | Baseline, 8 weeks, 16 weeks, 24 weeks.
  Fountas and Pinnell reading level

SECONDARY OUTCOMES:
Teacher perception of dance intervention | Baseline and 9 months.
  Survey of teachers knowledge and perception of dance in the classroom
Documented Student Behavior | 10 months.
  Referrals to principals office

CONTACTS AND LOCATIONS:
Overall Officials: Sarah DiPasquale, DPT, Principal Investigator — Skidmore College
Locations (1):
- Skidmore College, Saratoga Springs, New York, United States

IPD SHARING:
Plan to Share IPD: No
A linking list for students will be compiled by the school Principal, numerically coding each student into a password protected document. This student linking list will be kept on a locked district owned, password protected computer at the school, separate from this database. It will be kept solely on that computer hard drive so it will not be accessible to Principal at home. Neither the PI, nor any other Skidmore researchers will have access to this locked computer and therefore, will not have ability to gain access to this list in any capacity. Skidmore researchers will never have access to student names/identities.